CLINICAL TRIAL: NCT00488956
Title: Foot and Ankle Edema Post-Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H07-00540
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Foot and Ankle Edema
Keywords: foot; ankle; edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Some women develop swollen feet and ankles after a cesarean delivery. These women will often complain that their shoes are too tight and their feet may become numb or they may have some tingling in their feet.

Currently we do not know for sure that foot swelling occurs after a cesarean delivery and if it does what the cause is.

If we find that feet do swell after a cesarean delivery we may be able to suggest a cause. This may in the future prevent women developing excessive foot swelling.

We aim to investigate whether the size and shape of women's ankles do change following an elective cesarean delivery. We plan to investigate, if possible, the cause of any foot swelling after a cesarean whether it be the volume of intra venous fluids or oxytocin use.

DETAILED DESCRIPTION:
Pregnant women booked for an elective Cesarean delivery will be recruited into the study. Their foot volumes, based on volumetry, and foot and ankle circumferences will be measured prior to administration of IV fluids and then at 24 and 48 hours post delivery. They will also be questioned about their feet with regards to swelling, any symptoms of edema, and their mobility in the preceding two hours. Total fluid balance for the first 24 hours post delivery will be calculated, using the estimated blood loss in the OR, urine output, IV hydration and oral intake. The amount of oxytocin used will also be recorded. The parturient will be asked to fill in a form indicating the amount of oral fluid consumed in the first 24 hours post delivery. Information in the anaesthetic technique, height of block, use of vasopressors etc will be collected retrospectively from the anesthetic chart.

To reduce the chance of the caregivers altering their practice during the study, the attending anesthesiologist for the elective cesarean delivery will be unaware of the subject's participation in the study so that the IV fluids he or she gives will be as close to real practice as possible.

Current practice for IV start and infusion in the surgical daycare area will be used during the study period without modification.

Validation and reproducibility will also be investigated. Each investigator will measure the volume and circumference of the same limb 10 times and inter and intra tester reliability will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a singleton pregnancy;
2. Undergoing an elective CD under regional anesthesia (spinal or combined spinal epidural (CSE);
3. Normotensive; and
4. At least 37 weeks gestation

Exclusion Criteria:

1. Reasons for potential excessive blood loss (e.g. placenta previa);
2. Reasons for potential uterine atony and above average use of oxytocin (e.g. multiple pregnancies, polyhydramnios);
3. Non lower segment uterine incision;
4. Renal or cardiac disease;
5. Use of diuretics; or
6. Open wounds on the right foot and ankle.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women booked for an elective Cesarean delivery will be recruited into the study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roanne Preston, MD, Principal Investigator — University of British Columbia; Elizabeth Drake, MD, Study Director — University of British Columbia; Joanne Douglas, MD, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada